CLINICAL TRIAL: NCT00091897
Title: Efficacy of Rituximab in Patients With Stiff Person Syndrome With Anti-GAD Antibodies: A Randomized Placebo-Controlled Trial
Brief Title: Rituximab to Treat Stiff Person Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Marinos C. Dalakas, M.D./National Institute of Neurological Disorders and Stroke, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 040287; IND-BB: 11844, 04-N-0287
Record Dates: First submitted 2004-09-18; First posted 2004-09-20 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Stiff Person Syndrome
Keywords: RITUXAN; GABA; B Cells; Humanized Monoclonal Antibodies; GAD; Stiff Person Syndrome; SPS
MeSH Terms: conditions — Stiff-Person Syndrome | interventions — Rituximab

ARMS (1):
- Rituximab or placebo (Experimental): Rituximab or placebo is administered through intravenous access on day 1 and again on day 15 (+/- 2 days)
  Interventions: Drug: Rituximab; Drug: rituximab or placebo

INTERVENTIONS:
Drug: Rituximab
Drug: rituximab or placebo — A fixed dose of Rituximab or placebo 1GM on Day 1 and 1GM on day 15 (+/- 2 days)
  Other Names: Rituxan

SUMMARY:
This study will test whether rituximab (RITUXAN (Trademark)) can relieve symptoms of stiff person syndrome (SPS), a progressive disease that causes stiffness of the muscles and muscle spasms induced by unexpected noises, touches, or stressful events. People with SPS may have certain proteins in their blood called anti-GAD antibodies that may cause some of the symptoms of the disease. Rituximab, a drug approved to treat lymphomas, targets certain white blood cells that produce antibodies. This study will see if rituximab can also be effective in patients with SPS who have high anti-GAD antibodies.

Patients between 25 and 80 years of age with SPS may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood tests. Participants undergo the following tests and procedures:

* Rituximab or placebo treatment: Patients are randomly assigned to receive two infusions by vein of either rituximab or placebo (a look-alike solution with no active ingredient) 2 weeks apart. The infusions last from 3 to 4 hours, but may take as long as 16 hours if the rate must be slowed for any reason. Patients are followed monthly for up to 6 months and then every 2 months for up to 1 year after treatment.
* Medical history and interview, physical and neurological examinations: Patients are questioned about their vaccination history, medical, surgical, and psychiatric history, exposure to environmental toxins or viruses, and family and social history, including habits and employment.
* Blood drawing: Blood samples are collected before the two infusions and at all follow-up visits.
* Apheresis: For this procedure, which is used to collect white blood cells, blood is collected through a needle in an arm vein, similar to donating blood. The blood flows from the vein through a catheter (plastic tube) into a machine that separates it into its components by centrifugation (spinning). The white cells are removed and the rest of the blood (red cells, plasma and platelets) is returned to the body through a second needle in the other arm. The procedure takes about 60 to 90 minutes.
* Lumbar puncture (spinal tap): Lumbar puncture is done to sample a small amount of cerebrospinal fluid (CSF, the fluid that bathes the brain and spinal cord), for analysis. For this procedure, the patient is given a local anesthetic and a needle is inserted into the space between the bones in the lower back where the CSF circulates below the spinal cord. A small amount of fluid is withdrawn through the needle.

DETAILED DESCRIPTION:
This study will examine the safety, tolerability, and efficacy of the humanized monoclonal antibody Rituximab to induce a clinical and serological remission in patients with Stiff Person Syndrome (SPS) associated with high anti-GAD antibodies. Rituximab is a monoclonal antibody specific for the common B cell antigen CD20. Its administration depletes pre-B and mature B lymphocytes without altering neutrophils or hematopoietic stem cells. In humans with indolent B cell lymphomas, Rituximab can be safely administered, is well tolerated, promotes selective B cell depletion and lowers the serum IgG and IgM levels. Preliminary experience in some non-malignant antibody-mediated disorders has shown that Rituximab was beneficial in improving the patients' symptoms and reducing antibody level.

SPS is an antibody-mediated autoimmune disease affecting GABA-ergic transmission resulting in incapacitating stiffness and spasms. The anti-GAD antibodies are also produced intrathecally and it is believed to be responsible for the reduction of GABA level in serum and CSF. Although removal or modulation of serum antibodies by plasmapheresis or IVIg results in clinical improvement, a number of patients do not respond or their response is modest and short-lived, and remain with significant disability. The need for more effective therapy prompted us to conduct the present study to examine in a randomized trial if Rituximab is effective in patients with GAD-antibody-positive SPS.

Twenty-four patients will be randomized, in a double blind fashion, to receive placebo or Rituximab given at a fixed dose of 1 GM on Day 1and 1 GM on day 15 (plus or minus 2 days). The primary outcome will be based on measurements of stiffness using the Distribution of Stiffness Index. Secondary outcomes will be measured by the Heightened-Sensitivity Scales. The serum and CSF anti-GAD antibody titers, including intrathecal GAD-specific IgG synthesis, will be monitored before and after treatment. Clearance of GAD-reactive T cells will be also examined in the serum and CSF using T cell clones established from PBL and CSF. It is anticipated that the study will: a) provide a new, immune-based and target-oriented therapy for patients with Stiff Person Syndrome and b) examine the pathogenetic role of anti-GAD antibodies in the cause of the disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Stiff Person Syndrome with elevated anti-GAD antibody titers.

Between 25 to 80 years of age.

Willingness to stop IVIg therapy 6 weeks prior to Rituximab/Placebo treatment and for the remainder of the study. [If receiving IVIg, patients will be allowed to receive the ongoing non-immunosuppressive drugs used to treat SPS including Diazepam, Neurontin or Baclofen. The dose of these drugs will remain stable throughout the study and unchanged for 6 weeks prior to enrollment.]

Willingness and legal ability to give and sign informed study consent.

Willingness to travel to NIH for scheduled protocol studies and treatment.

Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.

Adequate bone marrow, renal, and liver function: ANC greater than 1000/mm(3), BUN/Cr in normal range for age.

Patients with Diabetes (Type II) will be allowed to participate because up to 40% of SPS patients have Diabetes.

Patients with a history of controlled epilepsy will be allowed to participate because up to 5% of SPS patients have mild epilepsy which is easily controlled.

EXCLUSION CRITERIA:

Immunosuppressive drug therapy for SPS at the time of or 6 weeks prior to enrollment and for the remainder of the study. Specifically, candidates may not be taking prednisone, cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, anti-lymphocyte agents, cyclophosphamide, methotrexate, or other agents whose therapeutic effect is immunosuppressive.

Any medical or social condition that precludes follow-up visits.

Any active malignancy or any history of a hematogenous malignancy or lymphoma. Patients with primary, cutaneous basal cell or squamous cell cancers may be enrolled providing the lesions are treated prior to enrollment.

History of a coagulopathy or patients requiring anticoagulation.

Any history of cardiac insufficiency, major vascular disease, or symptomatic coronary artery disease. Patients with cardiomyopathy grade III or IV by the New York Heart Classification will be excluded from this study.

Systemic edema or pulmonary edema.

Chronic and severe symptomatic hypotension (SBP less than 100 mmHg).

Chronic liver disease or alcoholism.

Any condition, including active infections, that would likely increase the risk of protocol participation or confuse the understanding of the data.

Pregnancy. Serum pregnancy test will be performed and must be negative in all women of childbearing potential enrolled in the study.

History of active psychiatric disorder that may interfere with participation in the study.

LABORATORY EXCLUSION CRITERIA (AT SCREENING):

Hemoglobin: less than 7.0 gm/dL.

Platelets: less than 100,000/mm.

AST or ALT greater than 2.5 x Upper Limit of Normal unless related to primary disease.

Positive Hepatitis B or C serology (Hep Surface antigen and Hep C hepatitis C antibody).

Positive HIV.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-09; Primary Completion 2007-07 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy, safety of the chimeric monoclonal antibody Rituximab to deplete B lymphocytes in patients with Stiff Person Syndrome with high anti-GAD antibodies. | 2 Years

SECONDARY OUTCOMES:
The Heightened Sensitivity Scale will be used as a secondary outcome measure. | 2 Years

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dalakas MC, Fujii M, Li M, McElroy B. The clinical spectrum of anti-GAD antibody-positive patients with stiff-person syndrome. Neurology. 2000 Nov 28;55(10):1531-5. doi: 10.1212/wnl.55.10.1531. PMID 11094109
- [Background] Dalakas MC, Li M, Fujii M, Jacobowitz DM. Stiff person syndrome: quantification, specificity, and intrathecal synthesis of GAD65 antibodies. Neurology. 2001 Sep 11;57(5):780-4. doi: 10.1212/wnl.57.5.780. PMID 11552003
- [Background] Levy LM, Dalakas MC, Floeter MK. The stiff-person syndrome: an autoimmune disorder affecting neurotransmission of gamma-aminobutyric acid. Ann Intern Med. 1999 Oct 5;131(7):522-30. doi: 10.7326/0003-4819-131-7-199910050-00008. PMID 10507962